CLINICAL TRIAL: NCT06300632
Title: Geriatric Locomotive Syndrome Kinesiophobia, Physical Activity Level, Physical Performance, Fatigue, Cognitive Functions in Older Adults
Brief Title: Geriatric Locomotive Syndrome and Related Factors in Older Adults
Status: Completed | Type: Observational
Sponsor: Kırıkkale University (Other)
Responsible Party: Principal Investigator, Ayşe Abit Kocaman, Principal Investigator, Kırıkkale University
Other Study IDs: Geriatric Locomotive Syndrome
Record Dates: First submitted 2024-02-28; First posted 2024-03-08 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-04

CONDITIONS: Locomotive Syndrome

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- older adults: older adults Geriatric Locomotive Function Scale Tampa Kinesiophobia Scale Physical Activity Scale for the Elderly (PASE) Brief Physical Performance Battery Fatigue Severity Scale Montreal Cognitive Assessment Scale (MoCA)
  Interventions: Other: geriatric locomotive syndrome

INTERVENTIONS:
Other: geriatric locomotive syndrome — Elderly individuals will be included in the study. Before each elderly person starts the study, they will be informed about the content of the study and they will read and sign the consent form stating that they participate in the study voluntarily. Socio-demographic data (age, body mass index, and family history, fall history, ) of all individuals participating in the study will be recorded.Within the scope of the evaluation, locomotive syndrome evaluation will be made through a survey. Fear of movement will be evaluated with the Tampa kinesiophobia scale, your physical activity level with the physical activity scale for the elderly, your physical performance with the short physical performance battery, your fatigue level with the fatigue severity scale, and your cognitive functions with the Montreal Cognitive Assessment Scale.

SUMMARY:
It has been stated that the results of physical function and physical performance affecting locomotive syndrome in elderly individuals are controversial and studies are still needed. However, no studies have been found examining its relationship with the decrease in physical activity level, decline in cognitive functions, kinesiophobia (fear of movement) and fatigue seen in old age. Early detection of locomotive syndrome risk factors in elderly individuals will help prevent this condition, detect the risk of falling in elderly individuals and increase their quality of life. Based on these deficiencies, it is aimed to examine the relationship between locomotive syndrome and kinesiophobia, physical activity level, physical performance, fatigue and cognitive functions in elderly individuals.

DETAILED DESCRIPTION:
It has been reported that problems related to the musculoskeletal system, such as osteoarthritis, osteoporosis or spondylosis, increase with aging in elderly individuals. The Japanese Orthopedic Association (JOA) has defined this condition as locomotive syndrome (LS) in elderly individuals, as a condition of decreased mobility due to deterioration of locomotive organs. LS is a condition of reduced mobility due to deterioration of locomotive organs. It has been stated that the results of physical function and physical performance affecting locomotive syndrome in elderly individuals are controversial and studies are still needed. However, no studies have been found examining its relationship with the decrease in physical activity level, decline in cognitive functions, kinesiophobia (fear of movement) and fatigue seen in old age. Early detection of locomotive syndrome risk factors in elderly individuals will help prevent this condition, detect the risk of falling in elderly individuals and increase their quality of life. Based on these deficiencies, it is aimed to examine the relationship between locomotive syndrome and kinesiophobia, physical activity level, physical performance, fatigue and cognitive functions in elderly individuals.

ELIGIBILITY:
Inclusion Criteria:

Individuals aged 65 and over, Volunteering to participate in research No cooperation and communication problems (Mini Mental State Test score above 24)

Exclusion Criteria:

Individuals with neurological and orthopedic problems

* Uncontrolled hypertension
* Those with cardiac disease
* Those with cooperation and communication problems

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: At Kırıkkale University Faculty of Health Sciences, Department of Physiotherapy and Rehabilitation, all elderly individuals aged 65 and over who meet the inclusion and exclusion criteria and who volunteer to participate in the study will be collected by face-to-face interview using evaluation forms.
Sampling Method: Non-Probability Sample
Enrollment: 97 (Actual)
Dates: Start 2024-04-15 (Actual); Primary Completion 2024-10-11 (Actual); Study Completion 2024-10-11 (Actual)

PRIMARY OUTCOMES:
Geriatric Locomotive Function Scale | Day 1
  It consists of a survey of 25 items, and each item is rated between 0 and 4 points. The total score is the result of the sum of all items ranging from 0 to 100; the higher the score, the greater the physical impairment of the elderly, and 16 points is the cutoff point for locomotive syndrome
Two Step Test | Day 1
  Two-step testing involves measuring step length for two steps. Individuals are asked to take two steps as long as possible and the longest measurement is recorded
Stand Up Test | Day 1
  In the stand-up test, the height of the lowest stool at which the individual can stand up from a sitting position with both feet or one leg is recorded. Stools of four heights are used: 40 cm, 30 cm, 20 cm and 10 cm. If the individual manages to hold the final standing position for more than 3 seconds without needing to take any additional steps, they are judged to have completed the trial.
Tampa Kinesiophobia Scale | Day 1
  Individuals' fear of movement (kinesiophobia) will be evaluated with the Tampa Kinesiophobia Scale, consisting of 17 items.People receive a total score between 17-68 points. A high score on the scale indicates that the person has a high level of kinesiophobia, that is, the fear of movement.
Physical Activity Scale for the Elderly (PASE) | Day 1
  The PASE evaluates physical activity performed over a 1-week time frame. Participation in leisure activities, including walking outside the home, light, moderate, and strenuous sport and recreation, and muscle strengthening were recorded as never, seldom (1-2 days/week), sometimes (3-4 days/week), and often (5-7 days/week) performed. PASE score was stratifi ed in tertiles: 0 to 40 (sedentary), 41 to 90 (light physical activity) and more than 90 (moderate to intense activity).
Short Physical Performance Battery | Day 1
  It consists of 3 objective tests that evaluate lower body function. These; 2.44 meter walking, getting up from a chair and standing balance test
Fatigue Severity Scale | Day 1
  Fatigue Severity Scale (FSS) is a scale that evaluates fatigue and consists of 9 questions. Each item is scored between 0 and 7.
Montreal Cognitive Assessment Scale (MoCA) | Day 1
  The scale includes items that evaluate attention and concentration, executive functions, memory, language, visual and spatial skills, abstract thinking, calculation and orientation dimensions. The lowest score that can be obtained from the scale is 0 and the highest score is 30. A low score indicates decreased cognitive functions

CONTACTS AND LOCATIONS:
Overall Officials: Ayşe Abit Kocaman, Principal Investigator — Kırıkkale University
Locations (1):
- Ayşe Abit Kocaman, Kırıkkale, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Inanaga S, Hasegawa M, Kosuge M, Ichimura S, Morii T, Hosogane N. Relationship between the 25-question Geriatric Locomotive Function Scale and physical function in the elderly people. J Bone Miner Metab. 2023 Jul;41(4):550-556. doi: 10.1007/s00774-023-01427-w. Epub 2023 Apr 8. PMID 37029834